CLINICAL TRIAL: NCT04694924
Title: Promoting Quality of Care: a Prospective Cohort Study of Localized and Locally Advanced Prostate Cancer Patients
Brief Title: Prospective Prostate Cancer and Patient-reported Outcomes Registry
Acronym: Prosquare
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: AZ Sint-Jan AV (Other); General Hospital Groeninge (Other); AZ Sint-Blasius Dendermonde (Unknown)
Responsible Party: Sponsor
Other Study IDs: S63359
Record Dates: First submitted 2020-12-24; First posted 2021-01-05 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate; Locally Advanced Prostate Carcinoma; Locally Advanced Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Localized and locally advanced prostate cancer: Localized prostate cancer (cT1a-T2c N0 M0) refers to the clinical condition where cancer is confined to the prostate gland, in the absence of lymph node invasion or metastases. Locally advanced refers to the extension of the tumor beyond the capsule of the prostate (cT3-T4) or the clinical presence of nodal invasion (cN+), without metastases.
  Interventions: Other: standard of care

INTERVENTIONS:
Other: standard of care — No other procedures than those performed during the usual care for prostate cancer patients will be done. No study medication will be provided as part of participation.
  Clinical outcomes will be reported via predefined electronic forms, integrated into the electronic health record (EHR). Patient-reported outcomes will be collected electronically.
  All treatment decisions will be made at the discretion of the investigator or treating physician.

SUMMARY:
This study aims to evaluate the use of a digital solution, integrated into the electronic health record, for prospective and structured reporting of clinical and patient-reported outcomes for patients diagnosed with localized or locally advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed diagnosis of localized or locally advanced prostate cancer
* Being able to speak, read and understand Dutch, French, or English
* Each patient (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he understands the purpose of, and is willing to participate in the study.

Exclusion Criteria:

* Patients with prior treatment for prostate malignancies will be excluded.
* Dementia, mental alteration, or psychiatric pathology that can compromise informed consent from the patient and/ or adherence to the protocol and the monitoring of the trial
* Patients who cannot submit themselves to following the protocol for psychological reasons, social, family, or geographical.
* Persons deprived of liberty or under guardianship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with newly diagnosed histologically proven localized and locally advanced prostate cancer referred to one of the participating sites will be eligible to be enrolled in the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of systematically reporting a standardized set of predefined clinical parameters | up to 10 years after diagnosis
  The proportion of patients who are enrolled in the registry over the total localized and locally advanced prostate cancer patients
Assessment of systematically collecting a predefined set of patient-reported outcomes | up to 10 years after diagnosis
  The proportion of patients who completed all questionnaires over the total of questionnaires send.

SECONDARY OUTCOMES:
Occurence of disease recurrence/progression | up to 10 years after diagnosis
  Biochemical prostate specific antigen (PSA) recurrence/progression and recurrence/progression based on medical imaging
General quality of life | at diagnosis, 6 months, 1 year, and annually up to 10 years after diagnosis
  Assessment of health-related quality of life in prostate cancer patients. Measured by EORTC Quality of Life Questionnaire C30 (QLQ-C30). The EORTC QLQ-C30 is a generic QoL questionnaire designed to cover issues important to all cancer patients
Prostate cancer specific quality of life | at diagnosis, 6 months, 1 year, and annually up to 10 years after diagnosis
  Measured by Extended Prostate cancer Index Composite 26 (EPIC26). EPIC-26 is a validated instrument that measures the quality of life across 5 disease-specific domains: urinary incontinence, urinary obstruction and irritation, bowel-related symptoms, sexual dysfunction, and hormonal symptoms.
Overall Survival (OS) | up to 10 years after diagnosis
  Overall survival is defined as the time from enrollment to date of death due to any cause.
Prostate Cancer (PC)-related Mortality (PM) | up to 10 years after diagnosis
  PC-related mortality is the death due to prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Everaerts, MD, PhD, Principal Investigator — UZ Leuven / KU Leuven
Locations (4):
- Belgium (4):
  - AZ Sint-Blasius, Dendermonde, Oost-Vlaanderen
  - University Hospitals Leuven, Leuven, Vlaams-Brabant
  - AZ Sint-Jan Brugge, Bruges, West-Vlaanderen
  - AZ Groeninge Kortrijk, Kortrijk, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: Undecided